CLINICAL TRIAL: NCT02600832
Title: Alcohol Approach Bias Modification to Decrease Problem Drinking and Impulsivity in Veterans With AUD: A Pilot Study
Brief Title: AABM to Decrease Problem Drinking and Impulsivity in Veterans With AUD: A Pilot Study
Acronym: AABM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24034
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2018-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AABM Training (Experimental): Immediately following screening, patients will be randomly assigned to receive 9 sessions of real AABM training (16 subjects each) taking place over three weeks.
  Interventions: Behavioral: AABM Training
- Sham Training (Sham Comparator): Immediately following screening, patients will be randomly assigned to receive 9 sessions of sham training (16 subjects each) taking place over three weeks.
  Interventions: Behavioral: Sham Training

INTERVENTIONS:
Behavioral: AABM Training — The investigators will use a training version of the Alcohol Approach-Avoidance Task (AAT), in which patients are asked to respond to the format of presented pictures, irrespective of the pictures' content. Pushing a presented picture away will decrease picture size, whereas pulling a picture closer will increase size. There are 2 categories of pictures; 20 different alcoholic and 20 different non-alcoholic beverages. Training effect is achieved by presenting alcohol pictures in push format only and non-alcoholic drinks in pull format only. Two hundred training trials are presented per session.
  Other Names: AABM
  Arms: AABM Training
Behavioral: Sham Training — Sham training is identical to AABM training, except pictures are presented randomly in both formats.
  Arms: Sham Training

SUMMARY:
The proposed study is a pilot prospective, parallel groups, randomized, double blind, sham training-controlled, 9-session (over 3 weeks) clinical trial of AABM in 32 male and female veterans entering treatment for AUD at the VA Medical Center at San Francisco, California, between ages 18-65. The study consists of screening, 3-week AABM training, Week-4 post-test, and Week-12 follow-up. Assessment of inhibitory control, alcohol approach bias and craving will be administered at baseline and Week-4. Immediately following screening, patients will be randomly assigned to receive 9 sessions of real or sham AABM training (16 subjects each) taking place over three weeks. Following the 3 weeks of training, patients will complete a Week-4 post-test which includes assessment of alcohol approach bias, inhibitory control, and craving and a Week-12 follow-up assessing drinking behavior.

DETAILED DESCRIPTION:
The overall goal of the proposed project is to improve the treatment of veterans who consume alcohol at hazardous or harmful levels. We will conduct a pilot controlled clinical trial to assess the feasibility and acceptability of implementing an Alcohol Approach Bias Modification (AABM) task in veterans seeking outpatient treatment for alcohol use disorder (AUD). The investigators will also explore the efficacy of AABM to reduce alcohol use and enhance executive function. The proposed study is designed to test AABM as a novel, acceptable, safe, low-cost intervention to augment and boost the efficacy of standard outpatient treatment for reducing alcohol use and simultaneously improving executive function in veterans with AUD.

The proposed project will pursue three primary aims in veterans with an AUD who are drinking alcohol at hazardous or harmful levels: 1) Establish the feasibility of enrolling and retaining veterans with AUD for a 3-week randomized trial of AABM; 2) Obtain preliminary assessment of the efficacy of AABM treatment to decrease alcohol approach bias and alcohol use; 3) Obtain preliminary assessment of the efficacy of AABM treatment to improve neurocognitive functioning domains that typically show deficits in AUD populations. To achieve these aims, we will conduct pilot prospective, parallel groups, randomized, double blind, sham training-controlled, 9-session (over 3 weeks) clinical trial of AABM in 32 male and female veterans entering treatment for AUD at the San Francisco VA Medical Center. We expect that this study will provide empirical data for recruitment, attrition and effect size estimation for a future randomized trial to definitively test that AABM reduces alcohol use and improves executive function in veterans with AUD. Moreover, findings from the proposed project are expected to improve the care of veterans with AUD, and by extension, to aid families and communities affected by the sequelae of these problems.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female veterans eligible for VA services.
2. Ages 18-65
3. Must meet criteria for current (not in remission) AUD using the Diagnostic Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
4. Must report "at-risk" or "heavy" drinking by NIH/NIAAA (National Institute on Health/National Institute on Alcohol Abuse and Alcoholism) criteria (>3 drinks/day or >7/week for women; >4 drinks/day or >14/week for men) for at least one week in the last 90 days.
5. Must express a desire to reduce, stop or abstain from alcohol use.
6. Must be enrolled in AUD treatment at the San Francisco Veterans Affairs Health Care System.

Exclusion Criteria:

1. Psychotic disorders, bipolar disorder, dementia, or other psychiatric or medical condition judged to be unstable.
2. Concurrent participation in another AUD treatment study.
3. Needing acute medical detoxification from alcohol based on a score ≥ 12 on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD).
4. Subjects legally mandated to participate in an alcohol treatment program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01; Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
retainment | 4 weeks
  Number of participants completing the 9 sessions of AABM or sham training divided by the total number of participants randomized to start AABM or sham training.

SECONDARY OUTCOMES:
Drinks per week (DPW) | 4 weeks
  Number of standard alcohol drinks per week.
Heavy Drinking Days Per Week (HDD) | 4 weeks
  Total number of heavy drinking days per week as defined by NIAAA criteria (>3 drinks/day for women; >4 drinks/day for men).

OTHER OUTCOMES:
Executive Function | 4 weeks
  z-score of executive function domains.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Medical Center San Francisco, San Francisco, California, United States